CLINICAL TRIAL: NCT02344160
Title: A Prospective, Multi-center Consecutive Series Study of Subjects Treated With the REDAPT™ Revision Femoral System
Brief Title: REDAPT Revision System Study to Assess 5 Year Revision Rate & up to 10 Year Revision Rate and Safety and Effectiveness
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit subjects
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-4538-02
Record Dates: First submitted 2015-01-14; First posted 2015-01-22 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Total Hip Arthroplasty (THA)
Keywords: Total Hip Arthroplasty; THA
MeSH Terms: interventions — Phlebotomy; Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Phlebotomy — Phlebotomy will be performed at study follow up visits to obtain blood for metal ion analysis which will monitor levels for safety outcome measures
  Other Names: blood draw

SUMMARY:
The objective of the study is to demonstrate non-inferiority of stem revision rate in subjects implanted with the REDAPT™ System with a revision rate of less than 9.8% at the 5 year mark assuming an observed rate of 6.5% at 5 years. Additional data will be collected as outcomes of safety and effectiveness data up to 10 years post REDAPT revision surgery.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, consecutive series study of subjects treated with REDAPT™. The safety and effectiveness of the REDAPT™ revision stem will be assessed over a maximum of 5 years with additional follow up to 10 years to assess outcomes. The objective of this study is to establish if the REDAPT™ stem revision rate is less than 9.8% at 5 years with an observed rate from literature review of 6.5% at 5 year.

ELIGIBILITY:
Inclusion Criteria:

* Subject requires revision hip arthroplasty
* Subject requires subsequent revision of a joint replacement that involves the insertion, removal and/or replacement of a prosthesis or implant
* Subjects with inflammatory degenerative joint disease including rheumatoid arthritis, arthritis secondary to a variety of diseases and anomalies, and congenital dysplasia; non-inflammatory degenerative joint disease (NIDJD) or any of its composite diagnoses of osteoarthritis, avascular necrosis, traumatic arthritis, slipped capital epiphysis, fused hip, fracture of the pelvis, and diastrophic variant
* Treatments of nonunion, femoral neck fracture and trochanteric fractures of the proximal femur with head involvement that are unmanageable using other techniques
* Endoprosthesis, femoral osteotomy, or Girdlestone resection
* Subject is at least 18 years of age
* Subject is skeletally mature in Investigators judgment
* Subject is willing to consent to participate in the study
* Subject is in stable health and is free of or treated and stabilized for cardiac, pulmonary, hematological, infection, or other conditions that would pose excessive operative risk

Exclusion Criteria:

* Known allergies to any components of the devices
* Subject is entered in another investigational drug, biologic, or device study within 30 days of active study participation
* Subject is known to be at risk for lost to follow-up, or failure to return for scheduled visits
* Subject is facing current or impending incarceration
* Female subject is of child-bearing age and not using an approved method of contraception
* Mental or neurological conditions which could impair the subject's ability or willingness to comply with the study
* Physical conditions or activities which tend to place extreme loads on implants, e.g., Charcot joints, muscle deficiencies, multiple joint disabilities, etc.
* Skeletal immaturity
* Subject is severely overweight (BMI > 40)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 340 subjects
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Stem revision | 5 years with additional follow up to 10 years
  the primary outcome will be assessed by the incidence of stem revision

SECONDARY OUTCOMES:
Revision for any reason | 5 years with additional follow-up to 10 years
  Revision for any reason
Radiographic Measurements | post operatively with additional follow-up to 10 years
  radiographic measurements to assess linear radiolucencies and subsidence to assess safety and potential change over time.
Hip Disability and Osteoarthritis Outcome Score (HOOS) and Euro Group Questionnaire (EQ-5D) | At baseline and up to 10 year follow up
  Subject reported outcomes will be collected and scored over time to assess change over time from baseline to 10 year post REDAPT Revision surgery
Harris Hip Score | at baseline and follow up visits up to 10 year follow up post surgically
  Clinical evaluations to score and assess changes over time from baseline to 10 year follow up post REDAPT Revision surgery
Number of participants with Adverse Events | Adverse events will be collected and assessed as safety out come at each study visit up to 10 years post surgery
  Adverse events will be collected to monitor safety
Metal Ion measurement in whole blood | baseline and at each study visit up to 10 years following REDAPT REvison surgery.
  blood will be analysed for metal ion levels at baseline and each study visit up to 10 years to assess change in serum metal ion level over time.

CONTACTS AND LOCATIONS:
Overall Officials: James Waddell, MD, Principal Investigator — St. Michaels Hospital
Locations (1):
- Ran Schwarzkopf, Irvine, California, United States